CLINICAL TRIAL: NCT04018469
Title: Patterned Electric Dressing Effects on Open Wounds
Acronym: PED
Status: Withdrawn | Type: Observational
Why Stopped: not enough staff to execute study
Sponsor: Gayle Gordillo (Other)
Responsible Party: Sponsor-Investigator, Gayle Gordillo, Professor, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 1807454805
Record Dates: First submitted 2019-03-11; First posted 2019-07-12 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Amputation; Open Wound
Keywords: PED Wound Dressing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples With DNA — wound debrided tissue and tissue biopsy sample
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No Interventions — No Interventions

SUMMARY:
1. This study is a pilot feasibility study to determine treatment effects to estimate sample size for future studies that evaluate wound bacteria colonization.
2. The secondary objective of this study aims to observe the effect of PED on an open wound and its effects in wound bacteria colonization.

DETAILED DESCRIPTION:
This study is designed as a pilot study where 30 patients receiving a below the knee amputation with at least one open wound on the limb will be enrolled. Patients are identified through medical records. The patients will be selected based on inclusion and exclusion criteria through pre-screening through the Comprehensive Wound Center's Limb Preservation Program and wound physicians/providers at Indiana University. The decision of amputation is made independently of the study and is solely made by the patient and their physician/provider. The provider decides based on the severity of the limb's condition if/when the limb should be amputated and will schedule this surgery with the patient based on current clinical standard of care. Study participation is decided independent of clinical decision. Patients enrolled in the study will wear the Patterned Electric Dressing (PED) on the wound(s) for up to 3 weeks or until amputation, whichever comes first and will have up to a total of 4 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older
* Patients identified to be receiving a non-traumatic below the knee amputation within 3 weeks of enrollment
* The affected limb to be amputated must have at least one open wound

  * Wound(s) must be able to be covered by 3x3 dressing
* Subjects willing and able to provide informed consent

Exclusion Criteria:

* Pregnant women
* Prisoners
* Individuals lacking consent capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study 30 patients receiving a below the knee amputation with at least one open wound on the limb will be enrolled. Patients are identified through medical records. The patients will be selected based on inclusion and exclusion criteria through pre-screening through the Comprehensive Wound Center's Limb Preservation Program and wound physicians/providers at Indiana University. Patients enrolled in the study will wear the Patterned Electric Dressing (PED) on the wound(s) for up to 3 weeks or until amputation, whichever comes first and will have up to a total of 4 study visits.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Bacterial colonization & culture | 3 weeks or until amputation, whichever comes first
  Bacteria colonization (cultures results high, moderate, low or negative).
Necrotic tissue assessed through light microscopy of tissue biopsies | 3 weeks or until amputation, whichever comes first
  Hematoxylin and Eosin staining of tissue sections to measure extent of tissue necrosis at baseline and compared to tissue obtained at surgery after PED treatment.% necrotic tissue will be measured.

SECONDARY OUTCOMES:
Wound area measured before and after wound treatment | 3 weeks or until amputation, whichever comes first
  To determine the effect of PED on % wound closure based on wound measurements at baseline and end of PED treatment.
Bacterial biofilm through Scanning Electron Microscopy analysis | 3 weeks or until amputation, whichever comes first
  Perform scanning electron microscopy to detect bacterial biofilm (high, moderate, low or negative) before and after PED treatment.
Bacterial contamination assessed through Colony Forming Units | 3 weeks or until amputation, whichever comes first
  Colony forming units will be measured from tissue samples and dressings to quantitate bacterial contamination levels at baseline and after PED treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gordillo Gayle, MD, Principal Investigator — Indiana University
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Ammons MC, Ward LS, James GA. Anti-biofilm efficacy of a lactoferrin/xylitol wound hydrogel used in combination with silver wound dressings. Int Wound J. 2011 Jun;8(3):268-73. doi: 10.1111/j.1742-481X.2011.00781.x. Epub 2011 Apr 1. PMID 21457463
- [Background] Costerton JW, Stewart PS, Greenberg EP. Bacterial biofilms: a common cause of persistent infections. Science. 1999 May 21;284(5418):1318-22. doi: 10.1126/science.284.5418.1318. PMID 10334980
- [Background] Douglas LJ. Medical importance of biofilms in Candida infections. Rev Iberoam Micol. 2002 Sep;19(3):139-43. PMID 12825991
- [Background] Schachter B. Slimy business--the biotechnology of biofilms. Nat Biotechnol. 2003 Apr;21(4):361-5. doi: 10.1038/nbt0403-361. No abstract available. PMID 12665817